CLINICAL TRIAL: NCT00076635
Title: An Open-Label Study of the Safety of Subcutaneous Recombinant Interferon Gamma-1b in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: An Open-Label Study of the Safety of Interferon Gamma-1b in Patients With IPF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: program discontinued based on GIPF-007 results
Sponsor: InterMune (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIPF-006
Record Dates: First submitted 2004-01-28; First posted 2004-01-30 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Lung Disease
Keywords: Idiopathic; Pulmonary; Fibrosis; IPF; Lung; Actimmune; Interferon; Gamma; InterMune
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Lung Diseases; Fibrosis | interventions — interferon gamma-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Interferon gamma-1b — 200 mcg, SQ, 3x per week

SUMMARY:
Open-label therapy will be administered to up to 220 patients, following completion of either InterMune Protocol GIPF-002 Part B or Protocol GIPF-004, to assess the long-term safety of subcutaneous Interferon gamma-1b. The study duration will be 5 years.

DETAILED DESCRIPTION:
Open-label therapy will be administered subcutaneously. Patients enrolled will continue to receive Interferon gamma-1b therapy three times per week and will be evaluated at 6-week intervals. Patients not taking Interferon gamma-1b at enrollment will re-initiate therapy with subcutaneous Interferon gamma-1b under a dose-escalation scheme, reaching full dose after 2 weeks.

ELIGIBILITY:
Inclusion criteria:

* Enrollment in Protocol GIPF 002 Part B or GIPF-004
* Completion of the End of Treatment Visit in Protocol GIPF-002 Part B or the Study Completion Visit in GIPF-004
* Able to understand and sign a written informed consent form and comply with the requirements of the study

Exclusion criteria:

* pregnancy or lactation
* lack of adherence to either GIPF-002 or GIPF-004 study protocols and treatment regimens
* if Principal Investigator deems patient is unsuitable for study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2003-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
All adverse events up to the end of study | 3.5 years
Survival status at end of study | 3.5 years
Serum antibodies to Interferon gamma-1b after the last injection. | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: InterMune, Inc. 888-486-6411 — Medical Information
Locations (1):
- Intermune Inc, Brisbane, California, United States